CLINICAL TRIAL: NCT00489229
Title: Studies on Diabetic and Pre Diabetic Vascular Disease and the Effect of Selected Therapeutic Modalities on Associated Vasculopathy
Brief Title: To Investigate the Effect of Rosiglitazone and Ramipril on Pre-clinical Vasculopathy in Diabetes and IGT Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: ID: 305/PPSP/6112215
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2009-07-16 (Estimated); Status verified 2007-03

CONDITIONS: Diabetes; Impaired Glucose Tolerance
Keywords: Rosiglitazone; Ramipril; Impaired glucose tolerance; Arterial stiffness; Diabetic vasculopathy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance | interventions — Rosiglitazone; Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rosiglitazone
Drug: Ramipril

SUMMARY:
The aim is to examine whether pharmacological interventions with thiazolidinedione and angiotensin converting enzyme (ACE) inhibitors can reverse pre-clinical vasculopathy in newly diagnosed diabetic and IGT individuals.

DETAILED DESCRIPTION:
The burden of diabetic vasculopathy on the global population is enormous and ever growing. Besides the well-known microvascular complications in type 2 diabetes (T2DM), there is a growing epidemic of macrovascular complications. People with T2DM have a higher risk of death from cardiovascular (CV) diseases than persons without diabetes. Like diabetes, impaired glucose tolerance (IGT) individuals also have associated risk of developing macrovascular complications. This calls for an early detection and intervention in patients with T2DM as well as IGT, not only to delay progression of IGT to T2DM but also to treat early macrovascular diseases in both groups. The traditional therapeutic approaches of T2DM emphasise on glycaemic control, which limits microvascular diseases but lacks an established benefit in macrovascular diseases. Type 2 diabetes is a metabolic disorder characterised by dyslipidaemia, hypertension, and hypercoagulability in addition to hyperglycaemia and hyperinsulinaemia. Each of these abnormalities plays an important role in diabetic vasculopathy and provides targets for therapy. Understanding the mechanisms of diabetic vasculopathy and instituting therapy guided by emerging evidences would improve outcomes in patients with T2DM and IGT.

In recent years, special attention has been devoted to both thiazolidinediones (TZDs) and angiotensin converting enzyme (ACE) inhibitors when TRIPOD study demonstrated that troglitazone may reduce the rate of progression to diabetes in women diagnosed with gestational diabetes and HOPE Study showed that ramipril may delay the onset of diabetes. The TZDs are novel insulin-sensitising antidiabetic agents, which also have vasculoprotective properties. Rosiglitazone, one of the members of TZD family, improves insulin sensitivity and may have a beta cell cytoprotective effect. The ACE inhibitors reduce both microvascular and macrovascular complications in diabetes and appear to improve insulin sensitivity and glucose metabolism. Ramipril, an ACE inhibitor, has direct effects on the renin-angiotensin-kallikrein system and may play an important role in the prevention of diabetes through effects on beta cell and by vascular and metabolic effects on muscle that may amplify the effects of insulin. Previous studies showed that newly diagnosed untreated T2DM/IGT and hypertensive Malay patients had early manifestations of preclinical vasculopathy and potentially increased risk for development of macrovascular diseases. The aim of this study is to investigate whether pharmacological interventions with rosiglitazone and ramipril can reverse pre-clinical vasculopathy in newly diagnosed untreated T2DM and IGT patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed untreated T2DM patients
* Newly diagnosed untreated IGT patients
* Normoglycaemic individuals
* Age: 30-65 years
* Blood Pressure <140/90 mmHg.

Exclusion Criteria:

* Patients with T2DM
* Hypertension (>140/90 mmHg)
* Microvascular and/or macrovascular complications of diabetes
* Severe hyperlipidaemia (>7.8 mmol/L)
* Smokers
* Obese people (BMI>30 Kg/m2)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2002-10; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Measuring arterial stiffness (pulse wave velocity and augmentation index) | One year

SECONDARY OUTCOMES:
Measuring fasting blood sugar and 2 hours post prandial sugars, fasting insulin level, HbA1c, and total cholesterol level. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Rashid A Rahman, MRCP, PhD, Study Director — Universiti Sains Malaysia
Locations (1):
- School of Medical Sciences, University Sains Malaysai, Kota Bharu, Kelantan, Malaysia

REFERENCES:
- [Derived] Rahman S, Ismail AA, Ismail SB, Naing NN, Rahman AR. Effect of rosiglitazone and ramipril on macrovasculopathy in patients with type 2 diabetes: needs longer treatment and/or higher doses? Clin Pharmacol. 2010;2:83-7. doi: 10.2147/CPAA.S8863. Epub 2010 Apr 20. PMID 22291490